CLINICAL TRIAL: NCT06194084
Title: Precision Nutrition - Impacts of Durian Consumption on Human Microbiome and Metabolome in Healthy Staff Volunteers From SingHealth
Brief Title: Impacts of Durian Consumption on Human Microbiome and Metabolome in Healthy Staff Volunteers
Acronym: DURIOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DURIOME
Record Dates: First submitted 2023-11-23; First posted 2024-01-08 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Diet, Food and Nutrition
Keywords: Precision Nutrition; Durian; Gut Microbiome; Metabolome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention - durian pulp. (Experimental): Two-sequence of doses (100 g and 200 g) of durian pulp.
  Interventions: Other: Two-sequence of durian pulp doses (100 g and 200 g)

INTERVENTIONS:
Other: Two-sequence of durian pulp doses (100 g and 200 g) — Participants first go through an initial washout maintaining a low-fiber diet for 14 days. After washout, participants will be instructed to consume 100 grams of durian pulp every day following their breakfast or dinner for 1 week. Participants will then continue to consume 200 grams of durian pulp every day during the 2nd week of intervention and then will go through another washout for 2 weeks.

SUMMARY:
This clinical study investigates the impacts of daily durian consumption on gut microbiota, gut microbial metabolites, and host metabolome in healthy individuals.

DETAILED DESCRIPTION:
Participants will go through an initial washout maintaining a low-fiber diet for 14 days. After washout, participants will be instructed to consume 100 grams of durian pulp every day following their breakfast or dinner for 1 week. Participants will then continue to consume 200 grams of durian pulp every day during the 2nd week of intervention and then will go through another washout for 2 weeks. During the intervention period, participants will be informed to maintain low-fiber diet. All participants will be required to note down their stool consistency and stool frequency and 3-days dietary records. Stool and blood samples will be collected at 4 time points during the study period (baseline, 1-week of intervention, 2-weeks of intervention and 2-weeks washout) and will be stored at -80 °C until analysis.

The first outcomes of this study will provide insights into the interplay between durian consumption, gut microbiome, and host metabolome, as well as whether durian consumption can improve the clinical parameters (plasma glucose levels, lipid profiles and HbA1c levels) of healthy subjects. The interplay between diets, gut microbiome, host metabolome and genetic polymorphism data in healthy population will lay the groundwork to develop the precision nutrition strategy based on our regional food. These findings have potential to improve the health and well-being of the communities in our region.

ELIGIBILITY:
Inclusion Criteria:

1. Male and/or female subjects between the ages of 21 and 60 years, inclusive
2. Willing and able to provide written informed consent
3. Must be in generally good health with clinically insignificant screening results (Fasting plasma glucose level & Lipid profile), as determined by the Investigator
4. Agrees to consume durian for 2 weeks
5. Agrees to maintain a low-fiber diet during the intervention
6. Have not received any antibiotics therapy, consumed prebiotics, probiotics, symbiotic /vitamin supplement, and/or TCM for at least 1 month before the start of the study
7. Have not received any medical treatment that would impact on intestinal microbiota at least 6 months before the start of the study or during the study
8. Recent COVID-19 vaccination received or infection with COVID-19 at least 2 months ago

Exclusion Criteria:

1. Known or suspected sensitivity/allergy to durian
2. Multiple food/drug allergies
3. Smoker
4. History or presence of current metabolic conditions and gastrointestinal diseases
5. Diagnosed with Inflammatory Bowel Disease (IBD) or significant liver enzyme abnormality
6. Presence of current haemorrhoids or piles causing rectal bleeding when passing stool
7. Pregnant, breastfeeding or intending to conceive during study period

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Fasted Blood Glucose | Baseline, 1 week after Intervention (100gm of durian consumption), 2 weeks after Intervention (200gm of durian consumption), Post-Intervention Wash-out (2 weeks after intervention).
  Changes in Fasted Blood Glucose (mg/dL), before & after Durian intervention.
HbA1C | Baseline, 1 week after Intervention (100gm of durian consumption), 2 weeks after Intervention (200gm of durian consumption), Post-Intervention Wash-out (2 weeks after intervention).
  Changes in HbA1C (%) before & after Durian intervention.
Total Cholesterol | Baseline, 1 week after Intervention (100gm of durian consumption), 2 weeks after Intervention (200gm of durian consumption), Post-Intervention Wash-out (2 weeks after intervention).
  Changes in Total Cholesterol (mg/dL) before & after Durian Intervention.
HDL Cholesterol | Baseline, 1 week after Intervention (100gm of durian consumption), 2 weeks after Intervention (200gm of durian consumption), Post-Intervention Wash-out (2 weeks after intervention).
  Changes in HDL Cholesterol (mg/dL) before & after Durian intervention.
LDL Cholesterol | Baseline, 1 week after Intervention (100gm of durian consumption), 2 weeks after Intervention (200gm of durian consumption), Post-Intervention Wash-out (2 weeks after intervention).
  Changes in LDL Cholesterol (mg/dL) before & after Durian intervention.
Cholesterol/HDL Ratio | Baseline, 1 week after Intervention (100gm of durian consumption), 2 weeks after Intervention (200gm of durian consumption), Post-Intervention Wash-out (2 weeks after intervention).
  Changes in Cholesterol/HDL ratio before & after Durian intervention.
Triglycerides | Baseline, 1 week after Intervention (100gm of durian consumption), 2 weeks after Intervention (200gm of durian consumption), Post-Intervention Wash-out (2 weeks after intervention).
  Changes in Triglycerides (mg/dL) before & after Durian intervention.
Carbohydrates | Baseline, 1 week after Intervention (100gm of durian consumption), 2 weeks after Intervention (200gm of durian consumption), Post-Intervention Wash-out (2 weeks after intervention).
  Food record for carbohydrate intake.
Protein | Baseline, 1 week after Intervention (100gm of durian consumption), 2 weeks after Intervention (200gm of durian consumption), Post-Intervention Wash-out (2 weeks after intervention).
  Food record for protein intake.
Fats | Baseline, 1 week after Intervention (100gm of durian consumption), 2 weeks after Intervention (200gm of durian consumption), Post-Intervention Wash-out (2 weeks after intervention).
  Food record for fat intake.
Dietary Fibre | Baseline, 1 week after Intervention (100gm of durian consumption), 2 weeks after Intervention (200gm of durian consumption), Post-Intervention Wash-out (2 weeks after intervention).
  Food record for dietary fibre intake.
Cholesterol | Baseline, 1 week after Intervention (100gm of durian consumption), 2 weeks after Intervention (200gm of durian consumption), Post-Intervention Wash-out (2 weeks after intervention).
  Food record for cholesterol intake.
Sodium | Baseline, 1 week after Intervention (100gm of durian consumption), 2 weeks after Intervention (200gm of durian consumption), Post-Intervention Wash-out (2 weeks after intervention).
  Food record for sodium intake.
Sugar | Baseline, 1 week after Intervention (100gm of durian consumption), 2 weeks after Intervention (200gm of durian consumption), Post-Intervention Wash-out (2 weeks after intervention).
  Food record for sugar intake.

SECONDARY OUTCOMES:
Changes in gut microbiome composition before and after Intervention. | Baseline, 1 week after Intervention (100gm of durian consumption), 2 weeks after Intervention (200gm of durian consumption), Post-Intervention Wash-out (2 weeks after intervention).
  The effect of intervention on alpha and beta diversity of the fecal microbial community will be evaluated by 16s sequencing (using illumina MiSeq platforms) of feal bacterial DNA at baseline and after each intervention period.
Changes in metabolomes before and after Intervention. | Baseline, 1 week after Intervention (100gm of durian consumption), 2 weeks after Intervention (200gm of durian consumption), Post-Intervention Wash-out (2 weeks after intervention).
  Changes in the plasma metabolomics will be evaluated via LC-QTOF-MS to identify the metabolomic markers at baseline and after each intervention period. Whereas changes in fecal microbial metabolomic will be determined via GC-QTOF-MS at baseline and after each intervention period.

OTHER OUTCOMES:
Plasma Samples obtained from 50 healthy participants form different multi-ethnicity (Malays, Chinese and Indians) will be genotyped using a custom single nucleotide polymorphism (SNP) genotyping array (Illumina OncoArray-500K Bead Chip). | Baseline.
  The association between the SNP in distinct ethnic groups and gut microbiome patterns will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Jason YS CHAN, MD, PhD, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided